CLINICAL TRIAL: NCT03545737
Title: Compare the Accuracy of the Distances Between the Midpoint of the Thyroid Cartilage to Suprasternal Notch Base on Body Surface Measurement Add the Distance Between Suprasternal Notch to Carina of Trachea According to Chest CT and Formula Base on Patient's Height as a Guide for the Intubation of a Left-sided Double-lumen Tube
Brief Title: Compare a New Method and Formula as a Guide for the Intubation of a Left-sided Double-lumen Tube
Status: Completed | Type: Observational
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Other Study IDs: 98776
Record Dates: First submitted 2018-05-15; First posted 2018-06-04 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Therapeutic Procedural Complication
MeSH Terms: interventions — Weights and Measures; Food, Formulated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Measurement: The distances between the midpoint of the thyroid cartilage to suprasternal notch base on body surface measurement add the distance between suprasternal notch to carina of trachea according to chest CT.
  Interventions: Other: Measurement
- Formula: The formula base on patient's height as a guide for the intubation of a Left-sided Double-lumen tube.
  The depth of intubation = 0.1977* height-4.2423
  Interventions: Other: Formula

INTERVENTIONS:
Other: Measurement — The distances between the midpoint of the thyroid cartilage to suprasternal notch base on body surface measurement add the distance between suprasternal notch to carina of trachea according to chest CT
  Groups: Measurement
Other: Formula — The formula base on patient's height as a guide for the intubation of a Left-sided Double-lumen tube
  Groups: Formula

SUMMARY:
One-lung ventilation (OLV) is required for the most of thoracic surgery to facilitate surgical visualization by collapsing the lung. The double-lumen tube (DLT) is the commonly used device for OLV. The objective of this study was to compare the accuracy of the distances between vocal cords to carina of trachea and formula base on patient's height as a guide for the intubation of a Left-sided Double-lumen tube

DETAILED DESCRIPTION:
In previous study, investigators found that the distances between vocal cords to carina of trachea was a useful predictive method for the intubation of a Left-sided Double-lumen tube. However in some hospitals preoperative chest CT scans not contain the vocal cords slice. So in this study investigators will compare the accuracy of the distances between the midpoint of the thyroid cartilage to suprasternal notch base on body surface measurement add the distance between suprasternal notch to carina of trachea according to chest CT and formula base on patient's height as a guide for the intubation of a Left-sided Double-lumen tube.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients undergoing elective left side thoracic surgery
2. Requiring a Uniblocker or DLT for one-lung ventilation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Age<18 or >70 years
  2. ASA>III; BMI>35kg/m2
  3. Without suspected tuberculosis or systemic infection
  4. Without severe cardiopulmonary disease, preoperative hoarseness and anticipated difficult airway
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
The incidence of the injuries of bronchi and carina | 1-3days
  The degree of bronchi and carina injuries: 1 clear; 2 a few petechiae; 3coalesced petechiae, hemorrhage, or ecchymosis; 4 erosion

SECONDARY OUTCOMES:
The incidence of dislodgement | 1 day
  The incidence of dislodgement after repositioning
The intubation time | 1-5min
  The intubation time (IT) was defined as the time from the anesthesiologist inserted the video laryngoscope between the teeth of patients until the double lumen-tube at the optimal position checked by Fiberoptic bronchoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- 中国, Qinhuangdao, Hebei, China